CLINICAL TRIAL: NCT00284986
Title: A Phase II Open Label Study to Evaluate the Safety and Efficacy of Prochymal (Ex-vivo Cultured Adult Human Mesenchymal Stem Cells) Infusion for the Salvage of Treatment-Refractory Acute GVHD Patients
Brief Title: Safety and Efficacy of Prochymal for the Salvage of Treatment-Refractory Acute GVHD Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Osiris 270-271
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2025-10-30 (Actual); Status verified 2023-04

CONDITIONS: Graft Versus Host Disease
Keywords: GVHD; Graft vs Host Disease; Graft versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — remestemcel-l

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PROCHYMAL™ (Experimental)
  Interventions: Drug: Prochymal

INTERVENTIONS:
Drug: Prochymal — Intravenous infusion of ex-vivo cultured adult human mesenchymal stem cells

SUMMARY:
This study is designed to evaluate the safety and efficacy of Prochymal® (Ex-vivo Cultured Adult Human Mesenchymal Stem Cells) in participants experiencing treatment-refractory acute GVHD, Grades III-IV, that is refractory to standard first-line therapies and at least one second-line therapy.

DETAILED DESCRIPTION:
Allogeneic HSCT is used in the treatment of a variety of hematological, myeloproliferative and lymphoproliferative disorders, and malignancies involving solid tumors. Participants receiving HSCT can develop a life-threatening condition called GVHD. GVHD occurs when donor T cells from the donor bone marrow recognize host cells as "foreign" and initiate an inflammatory immunological response. The standard of care for treatment of acute GVHD consists of intravenous delivery of methylprednisolone starting on Day 1 and continuation of either cyclosporine or tacrolimus. This regimen of steroids and immunosuppressive drugs may relieve symptoms of GVHD, but some participants are refractory to current standard of care treatment. For treatment-refractory participants with grades III-IV GVHD mortality is approximately 80%. A therapy that could effectively suppress the immunological response from GVHD and help repair the damaged tissue could significantly decrease the mortality rate from this disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 6 months to 70 years of age inclusive.
* If female and of childbearing age, participants must be non-pregnant, not breast-feeding, and use adequate contraception. Male participants must use adequate contraception.
* Participants must have Grade III-IV acute GVHD that has failed to respond to standard first and at least one second-line therapy. Biopsy for confirmation of both skin and gastrointestinal GVHD is not mandatory, but is recommended when feasible. Enrollment should not be delayed awaiting biopsy results.
* Participants must have minimal renal function as defined by: Calculated creatinine clearance (CrCl) of > 30 milliliters/minute (mL/min) using the Cockcroft-Gault equation.
* Participant must provide written informed consent and authorization for use and disclosure of protected health information (PHI).

Exclusion Criteria:

* Participant has uncontrolled alcohol or substance abuse within 6 months of treatment.
* Participant has any underlying or current medical or psychiatric condition that, in the opinion of the Investigator, would interfere with the evaluation of the participant (e.g., uncontrolled infection, right heart failure, pulmonary hypertension, etc.).
* Participant has a clinically significant, unstable arrhythmia.
* Participant has a known allergy to bovine or porcine products.
* Participant is unwilling to sign consent form for the long-term follow-up study, protocol 271.

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-11-18 (Actual); Primary Completion 2006-04-25 (Actual); Study Completion 2007-02-08 (Actual)

PRIMARY OUTCOMES:
Response by Day 28 | Day 28
  Responses included complete response (CR), partial response (PR), failure to respond. CR is defined as a complete resolution of graft-versus-host disease (GVHD). PR is defined as improvement in at least one organ by at least one full stage in the absence of progression in any other organ, or resolution of GVHD in at least one organ with a need for additional treatment because of abnormalities persisting in another organ. Failure to respond is defined as progression of GVHD.

SECONDARY OUTCOMES:
Improvement of GVHD by Day 28 in one or more organs involved with GVHD symptoms at day 1 | Day 1
Best stage of each involved organ by Day 28 | Day 28
Time to improvement or resolution of GVHD in one or more organs | Up to approximately 12 months
Adverse events | Up to approximately 12 months
Infusional toxicity | Up to approximately 12 months
Overall relapse of underlying disease | Up to approximately 12 months
Overall survival | Up to approximately 12 months
Formation of ectopic tissue foci | Up to approximately 12 months
Incidence of infection | Up to approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher James, PA, Study Director — Mesoblast, Inc.
Locations (1):
- Duke University, Durham, North Carolina, United States